CLINICAL TRIAL: NCT01198353
Title: Study Evaluating Effectiveness of Ziprasidone Using the Overlapped Switching Strategy in Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Effectiveness of Ziprasidone for Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Han Yong Jung, Professor, Soonchunhyang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG-KOR-017-2009
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Ziprasidone; Switch; Metabolic syndrome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Metabolic Syndrome | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ziprasidone (Experimental): During the 12-week study period, patients were prescribed ziprasidone at 20 to 160 mg/day flexibly based on their effectiveness and tolerability. Fifty to one hundred percent of the past antipsychotic dose was maintained in the first week; during next 3 weeks, flexible dosing of 0-100% was used; then, ziprasidone was discontinued. This study included four visits: baseline, week 4, week 8, and week 12. Concomitant benzodiazepines (oral formula or injection) were allowed up to a dose of 4 mg of lorazepam-equivalents per day for anxiety and agitation.
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — 100% of the past antipsychotic dose will be maintained in week 1, using flexible dosing of 0-100% during next 3 weeks and then discontinued. Ziprasidone will be maintained with flexible dosing of 40-160mg/day during the study period.
  Other Names: Zeldox

SUMMARY:
This study is designed with the aim to evaluate the clinical effect of the overlapped switching to ziprasidone as well as the efficacy and safe metabolic profile of ziprasidone.

DETAILED DESCRIPTION:
Patients with schizophrenia or schizoaffective disorder were recruited in this 12-week, multicenter, non-comparative, open-label trial. Prior antipsychotics were allowed to be maintained for up to 4 weeks during the titration of ziprasidone. Efficacy was primarily measured using the 18-item Brief Psychotic Rating Scale (BPRS) at baseline, 4 weeks, 8 weeks, and 12 weeks. Efficacy was secondarily measured by the Clinical Global Impression - Severity (CGI-S) scale and the Global Assessment of Functioning (GAF) scale at each visit. Regarding the metabolic effects of switching to ziprasidone, weight, body mass index (BMI), waist-to-hip ratio (WHR), and lipid profile-including triglyceride (TG), high-density lipoprotein (HDL), low-density lipoprotein (LDL), and total cholesterol levels-were measured at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18-55 years treated with risperidone, olanzapine, amisulpride, quetiapine and typical antipsychotics.
* Both in- and outpatients who met Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for schizophrenia or schizoaffective disorder.
* Their primary psychiatric clinician determined that they would benefit from a change in their medications, either because of suboptimal efficacy or because of side effects.

Exclusion Criteria:

* Those who are treated with medications that prolong the QTc interval.
* Those who have any other axis I DSM-IV diagnoses.
* Those who have a history of substance abuse or dependence within 1 month.
* Those who have clinically significant abnormal laboratory values or any other abnormal baseline laboratory findings considered by psychiatrists to be indicative of conditions that might affect the study results.
* Those who have a past history of hypersensitivity or intolerance to ziprasidone.
* Those who have history of clozapine use within 1 month.
* Those who participated in clinical trials within 1 month before entering the study entry.
* Those who have used depot antipsychotics within one cycle before entering the study.
* Those who are pregnant or are breast feeding.
* Those who have a immediate risk of harming self or others or history of suicide attempts in the year before the screening precluded inclusion in the study.
* The patients unable/unlikely to comprehend/follow the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
A change in the Brief Psychotic Rating Scale (BPRS) | baseline and 12 weeks

SECONDARY OUTCOMES:
A change in the Lipid profile (Triglyceride, HDL, LDL, Total cholesterol) | baseline and 12 weeks
A change in the Body Mass Index (BMI) | baseline and 12 weeks
A change in the Waist-to-hip ratio | baseline and 12 weeks
UKU side effect rating scale - patient (UKU-SERS-Pat) | baseline
UKU side effect rating scale - patient (UKU-SERS-Pat) | 4 weeks
UKU side effect rating scale - patient (UKU-SERS-Pat) | 8 weeks
UKU side effect rating scale - patient (UKU-SERS-Pat) | 12 weeks
A change in the Clinical Global Impression (CGI) | Baseline and 12 weeks
A change in the Global Assessment of Functioning (GAF) | Baseline and 12 weeks
Blood chemistry tests including CBC, electrolyte, LFT, Nitrogen Elements, and protein | Baseline
Blood chemistry tests including CBC, electrolyte, LFT, Nitrogen Elements, and protein | 12 weeks
Urinalysis | Baseline
Urinalysis | 12 weeks
Electrocardiogram (ECG) | Baseline
Electrocardiogram (ECG) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Han Yong Jung, MD, PhD, Principal Investigator — DEPARTMENT OF PSYCHIATRY SOONCHUNHYANG UNIVERSITY BUCHEOMN HOSPITAL
Locations (6):
- South Korea (6):
  - Korea University Medical Center Ansan Hospital, Ansan, Gyeonggi-do
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Inha University Hospital, Incheon
  - Catholic University Our Lady of Mercy Hospital, Incheon
  - Korea University Medical Center Guro Hospital, Seoul
  - Kangnam Sacred Heart Hospital, Seoul

REFERENCES:
- [Background] Kudla D, Lambert M, Domin S, Kasper S, Naber D. Effectiveness, tolerability, and safety of ziprasidone in patients with schizophrenia or schizoaffective disorder: results of a multi-centre observational trial. Eur Psychiatry. 2007 Apr;22(3):195-202. doi: 10.1016/j.eurpsy.2006.06.004. Epub 2006 Nov 29. PMID 17140769
- [Background] Weiden PJ, Newcomer JW, Loebel AD, Yang R, Lebovitz HE. Long-term changes in weight and plasma lipids during maintenance treatment with ziprasidone. Neuropsychopharmacology. 2008 Apr;33(5):985-94. doi: 10.1038/sj.npp.1301482. Epub 2007 Jul 18. PMID 17637612
- [Background] Stip E, Zhornitsky S, Potvin S, Tourjman V. Switching from conventional antipsychotics to ziprasidone: a randomized, open-label comparison of regimen strategies. Prog Neuropsychopharmacol Biol Psychiatry. 2010 Aug 16;34(6):997-1000. doi: 10.1016/j.pnpbp.2010.05.010. Epub 2010 May 12. PMID 20470848
- [Background] Montes JM, Rodriguez JL, Balbo E, Sopelana P, Martin E, Soto JA, Delgado JF, Diez T, Villardaga I. Improvement in antipsychotic-related metabolic disturbances in patients with schizophrenia switched to ziprasidone. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Mar 30;31(2):383-8. doi: 10.1016/j.pnpbp.2006.10.002. Epub 2006 Nov 28. PMID 17129654
- [Background] Alptekin K, Hafez J, Brook S, Akkaya C, Tzebelikos E, Ucok A, El Tallawy H, Danaci AE, Lowe W, Karayal ON. Efficacy and tolerability of switching to ziprasidone from olanzapine, risperidone or haloperidol: an international, multicenter study. Int Clin Psychopharmacol. 2009 Sep;24(5):229-38. doi: 10.1097/YIC.0b013e32832c2624. PMID 19531959